CLINICAL TRIAL: NCT03845270
Title: Phase II Trial of Trastuzumab in Combination With Pertuzumab in Pretreated Patients With Non-small Cell Lung Cancer (NSCLC) Harboring a Her2 Mutation and Receiving Docetaxel
Brief Title: Her2-positive Lung Cancer Treated With Dedicated Drug
Acronym: R2D2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1703
Record Dates: First submitted 2019-02-14; First posted 2019-02-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Non Small Cell Lung Cancer Metastatic; Non Small Cell Lung Cancer Stage III; HER2 Gene Mutation
Keywords: IFCT; NSCLC; HER2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pertuzumab; Trastuzumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pertuzumab + trastuzumab + docetaxel (Experimental): Cycle 1 : D1 : pertuzumab 840 mg, D2 : trastuzumab 8 mg/kg + docetaxel 75 mg/m² Subsequent cycle : D1 : pertuzumab 420 mg + trastuzumab 6 mg/kg + docetaxel 75 mg/m²
  Interventions: Drug: pertuzumab + trastuzumab + docetaxel

INTERVENTIONS:
Drug: pertuzumab + trastuzumab + docetaxel — Cycle 1 : D1 : pertuzumab 840 mg, D2 : trastuzumab 8 mg/kg + docetaxel 75 mg/m² Subsequent cycle : D1 : pertuzumab 420 mg + trastuzumab 6 mg/kg + docetaxel 75 mg/m²

SUMMARY:
HER2 (erbB-2/neu) is a member of the erbB receptor tyrosine kinase family. ERBB2 gene which encodes human epidermal growth factor 2 (HER2) is a major proliferative driver activating downstream signaling through PI3K-AKT and MEK-ERK. HER2 overexpression or gene amplification is associated with sensitivity to trastuzumab and lapatinib in breast cancer. Among actual lung cancer biomarker, HER2 remains apart. HER2 involvement is known for a long time but clinical research has been stopped for many years since the first clinical trials in unselected patients were negative. Recently trastuzumab + pertuzumab + docetaxel has been tested for first-line treatment of HER2-positive metastatic breast cancer (CLEOPATRA trial). Analysis of the primary end point showed that patients who received pertuzumab, trastuzumab, and docetaxel (pertuzumab group) had a significantly longer median progression-free survival, as assessed by independent reviewers an did those who received placebo, trastuzumab, and docetaxel (control group) (hazard ratio favoring the pertuzumab group, 0.62). There is thus a strong rational for treating HER2 mutated lung cancer patient with these drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Patient having signed an informed consent form
2. Histologically or cytologically confirmed NSCLC (per 2015 8th edition TNM classification)
3. Not suitable for radiation, inoperable stage III or stage IV
4. HER2 exon 20 mutation or insertion among which: in-frame insertions in exon 20 between codons 775 and 881 including the 12bp insertion with a duplication / insertion of 4 amino acids (YVMA) at codon 775, the 3bp insertion with a complex insertion-substitution G776>VC and point mutations L755S and G776C. Other mutation/insertion should be discussed with IFCT. Analysis must be performed in INCa-labelled laboratories or platforms according to a validated procedure.
5. Prior treatment with at least one regimen of platinum-based chemotherapy with documented disease progression.

   Note: taxanes are allowed provided that no grade >2 associated adverse event occurred (except hematological toxicity).
6. Presence of at least one lesion that can be measured by CT scan (RECIST v1.1)
7. Age ≥ 18 years
8. Adequate organ function, as evidenced by the following laboratory results:

   ANC > 1500 cells/mm3 Platelet count > 100,000 cells/mm3 Hemoglobin > 9.0 g/dL Patients are allowed to receive transfused RBC to achieve this level. Total bilirubin ≤ 1.5 × ULN, except in patients with previously documented Gilbert's syndrome, in which case the direct bilirubin should be less than or equal to the ULN SGOT and SGPT ≤ 2.5 × ULN Alkaline phosphatase ≤ 2.5 × ULN, Alkaline phosphatase < 5×ULN and SGOT and SGPT < 5×ULN for patients with hepatic and/or bone metastases Clearance creatinine ≥ 30 mL/min INR and aPTT ≤ 1.5 x ULN This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
9. WHO performance index of 0, 1 or 2
10. LVEF ≥ 50%
11. Patient who is capable, according to the investigator, of complying with the study's requirements and restrictions
12. Estimated life expectancy > 3 months
13. A female is eligible to enter and participate in this study if she is of:

    Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has undergone:
    * Hysterectomy.
    * Bilateral oophorectomy (ovariectomy).
    * Bilateral tubal ligation.
    * Or who is post-menopausal:
    * Patients not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone value >40 mIU/mL and an estradiol value <40 pg/mL (<140 pmol/L).
    * Patients must discontinue HRT prior to study enrolment due to the potential for inhibition of cytochrome enzymes that metabolize estrogens and progestins. For most forms of HRT, at least 2 4 weeks must elapse between the cessation of HRT and determination of menopausal status; length of this interval depends on the type and dosage of HRT. If a female subject is determined not to be post-menopausal, they must use adequate contraception, as defined immediately below.

    Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception during the study and for at least 7 months after the last dose of investigational product. Contraceptive methods acceptable to IFCT, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:
    * A non-hormonal intrauterine device with a documented failure rate of less than 1% per year.
    * Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
    * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 7 months after the last dose of investigational product.
    * Two effective forms of non-hormonal contraception (condom with spermicidal jelly, foam suppository or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).

    Note: Oral contraceptives are not allowed.
14. Female patients who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 15 days following the last dose of study drug.
15. A male with a female partner of childbearing potential is eligible to enter and participate in the study if he uses a barrier method of contraception or abstinence during the study and for at least 7 months after the last dose of investigational product.
16. Patient will be eligible for inclusion in this study only if either affiliated to or a beneficiary of social security insurance.

Exclusion Criteria:

1. History of cancer except cancer dating from over two years ago and considered to be cured, appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma and stage I uterine cancer.
2. Any approved anti-cancer therapy ≤ 21 days before enrollment. Note: TKIs approved for the treatment of NSCLC must be discontinued ≥ 7 days prior to the first study treatment on Cycle 1, Day 1. (The baseline scan must be completed after discontinuation of TKIs).
3. Patients with concomitant EGFR, ALK, ROS1, MET, BRAF and KRAS mutation. Other molecular co-alterations should be discussed with IFCT before patient's enrollment.
4. Previous treatment with an anti-HER2 agent.
5. Any other investigational therapy ≤ 28 days before inclusion
6. Previous irradiation <14 days before enrollment.
7. Brain metastases that are symptomatic, or require any radiation, surgery, or corticosteroid therapy to control symptoms from brain metastases within 4 weeks before enrollment. Asymptomatic brain metastases with a fixed dose of steroids for at least 2 weeks are eligible.
8. Carcinomatous meningitis
9. History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab, pertuzumab or docetaxel or murine proteins or one of the excipients
10. Pregnancy and breast-feeding
11. Any evidence of severe or uncontrolled systemic disease. (E.g. unstable or uncompensated respiratory, cardiac, hepatic, or renal disease) or other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study.
12. Evidence of active pneumonitis during screening
13. Current unstable ventricular arrhythmia requiring treatment, history of symptomatic congestive heart failure (CHF; New York Heart Association [NYHA] Classes II-IV) and history of myocardial infarction or unstable angina within 6 months before enrollment.
14. Unresolved toxicity grade > 2 from previous anti-tumor treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Overall Response | [Time Frame: About 24 months]
  Proportion of patients with a confirmed complete response or partial response according to RECIST version 1.1

SECONDARY OUTCOMES:
Objective Response Rate | 6 weeks
  Percentage of patient with objective response rate with RECIST 1.1 as assessed by radiology review committee
Overall Survival | About 24 months
  Time from enrollment until death due to any cause
Progression-free survival | About 24 months
  Time from enrollment to first observation of progression (according to RECIST v1.1) or date of death (from any cause)
Duration of response | About 24 months
  Time from documentation of tumor response to disease progression.
Objective Response Rate | 6 weeks (confirmation needed at least after 4 weeks)
  Percentage of patient with objective response rate with RECIST 1.1 as assessed by investigators
Incidence, type and severity of non-serious and serious adverse event | About 24 months

OTHER OUTCOMES:
Correlation between OR, PFS, and HER2 mutation kinetic on cfDNA | About 24 months

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - Caen - CHU Côte de Nacre, Caen
  - Clermont-Ferrand - CHU, Clermont-Ferrand
  - CHI Créteil, Créteil
  - CHRU Grenoble, Grenoble
  - Centre Hospitalier - Pneumologie, Le Mans
  - Lyon - URCOT, Lyon
  - Hôpital Nord APHM, Marseille
  - Montpellier - CHRU, Montpellier
  - CHU de Nantes, Nantes
  - Nice CLCC, Nice
  - AP-HP Hopital Tenon - Pneumologie, Paris
  - AP-HP Hôpital Bichat, Paris
  - Rennes - CHU, Rennes
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mazieres J, Lafitte C, Ricordel C, Greillier L, Negre E, Zalcman G, Domblides C, Madelaine J, Bennouna J, Mascaux C, Moro-Sibilot D, Pinquie F, Cortot AB, Otto J, Cadranel J, Langlais A, Morin F, Westeel V, Besse B. Combination of Trastuzumab, Pertuzumab, and Docetaxel in Patients With Advanced Non-Small-Cell Lung Cancer Harboring HER2 Mutations: Results From the IFCT-1703 R2D2 Trial. J Clin Oncol. 2022 Mar 1;40(7):719-728. doi: 10.1200/JCO.21.01455. Epub 2022 Jan 24. PMID 35073148
- See also: IFCT website — https://www.ifct.fr/etudes-cliniques/148-ifct-1703